CLINICAL TRIAL: NCT06863116
Title: Peri-Implant Hypoxia as a Potential Barrier Against Ferroptotic Mechanisms During Peri-Implant Diseases
Brief Title: Analysis of HIF-1α, MDA, and GPX4 in Peri-Implant Crevicular Fluid
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Büşra Yılmaz, Professor, Ege University
Other Study IDs: 23-4.1T/14
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis; Hypoxia; Ferroptosis
Keywords: Peri-Implantitis; Peri-implant mucositis; Hypoxia; Ferroptosis; Lipid Peroxidation
MeSH Terms: conditions — Peri-Implantitis; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peri-implant crevicular fluid (PICF) samples were collected from study participants for biomarker analysis. No DNA extraction is planned from these samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peri-Implant Health: Participants with no clinical signs of peri-implant disease. These individuals exhibit healthy peri-implant soft tissues with no bleeding on probing (BOP), probing depth (PD) ≤ 4 mm, and no radiographic bone loss.
- Peri-Implant Mucositis: Participants diagnosed with peri-implant mucositis, characterized by bleeding on probing (BOP) and/or signs of inflammation (redness, swelling), but without radiographic bone loss beyond early remodeling.
- Peri-Implantitis: Participants diagnosed with peri-implantitis, defined by increased probing depth (PD > 5 mm), bleeding on probing (BOP) or suppuration, and radiographic evidence of bone loss beyond initial remodeling.

SUMMARY:
Peri-implant diseases, such as peri-implant mucositis and peri-implantitis, are inflammatory conditions that affect the tissues surrounding dental implants. If untreated, these diseases can lead to bone loss and implant failure. This study investigates whether low oxygen levels (hypoxia) in the peri-implant environment influence ferroptosis, a type of cell death associated with oxidative stress. The research focuses on three key biomarkers: hypoxia-inducible factor-1 alpha (HIF-1α), glutathione peroxidase-4 (GPX-4), and malondialdehyde (MDA).

A total of 45 participants with 62 dental implants were included in the study. They were divided into three groups: peri-implant health, peri-implant mucositis, and peri-implantitis. Peri-implant crevicular fluid (PICF) samples were collected, and the levels of HIF-1α, GPX-4, and MDA were measured using laboratory tests.

The study aims to determine whether hypoxia affects ferroptosis-related pathways by altering GPX-4 and MDA levels. Understanding these mechanisms could provide new insights into peri-implant disease progression and help develop improved treatment strategies.

DETAILED DESCRIPTION:
Peri-implant diseases are characterized by an inflammatory response leading to progressive bone loss around dental implants. While microbial biofilms and host immune responses contribute to disease progression, recent studies have suggested that programmed cell death pathways, including ferroptosis, may also play a role. Ferroptosis is an iron-dependent form of non-apoptotic cell death that is regulated by GPX-4, a key enzyme that prevents lipid peroxidation, and MDA, a biomarker of oxidative damage. Hypoxia, a common feature in peri-implant disease, is known to modulate oxidative stress and inflammatory responses through HIF-1α, but its role in ferroptosis remains unclear.

This cross-sectional study aims to evaluate the relationship between hypoxia and ferroptosis in peri-implant diseases by measuring the levels of HIF-1α, GPX-4, and MDA in peri-implant crevicular fluid (PICF). A total of 45 participants with 62 dental implants were included in the study, categorized into peri-implant health (PH), peri-implant mucositis (PM), and peri-implantitis (PP) groups. PICF samples were collected using standardized paper strips, and biomarker levels were quantified via enzyme-linked immunosorbent assay (ELISA). Statistical analyses, including Kruskal-Wallis and Spearman correlation tests, were performed to assess differences among groups and potential associations between biomarkers.

The findings demonstrated that MDA levels were significantly lower in the peri-implantitis and peri-implant mucositis groups compared to peri-implant health, while GPX-4 levels were elevated in peri-implant mucositis and decreased in peri-implantitis. HIF-1α levels showed no significant differences among groups, but a positive correlation was observed between HIF-1α and GPX-4, suggesting a potential interaction between hypoxia and ferroptotic regulation in peri-implant tissues. These results imply that hypoxic conditions in peri-implant diseases may inhibit ferroptosis by modulating GPX-4 activity and reducing lipid peroxidation.

The study provides novel insights into the pathophysiology of peri-implant diseases, suggesting that the peri-implant microenvironment may exhibit unique regulatory mechanisms affecting ferroptotic pathways. While these findings contribute to our understanding of peri-implant disease pathogenesis, further longitudinal studies are needed to establish causal relationships and explore potential therapeutic strategies targeting hypoxia-ferroptosis interactions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least one dental implant functioning for a minimum of one year.
* No history of systemic diseases.
* No periodontal treatments (surgical or non-surgical) in the past six months.
* No use of antibiotics or other medications within the past six months.

Exclusion Criteria:

* Systemic diseases, including but not limited to:

Diabetes mellitus Rheumatoid arthritis Cardiovascular disorders Immunological disorders Mucocutaneous diseases Contagious or communicable diseases

* Medication use, including:

Immunosuppressants Steroids Non-steroidal anti-inflammatory drugs (NSAIDs) Antiepileptics Calcium channel blockers Beta-blockers Anticoagulants Hormonal contraceptives Nutritional supplements

* Pregnant or lactating women.
* Use of orthodontic appliances or removable partial dentures.
* Poorly maintained implant-supported prostheses that may interfere with peri-implant crevicular fluid collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included individuals with at least one dental implant, recruited from the Department of Periodontology, Ege University, Faculty of Dentistry. Participants were selected based on specific eligibility criteria, ensuring that they had an implant functioning for at least one year and no history of systemic diseases or recent periodontal treatments. The study population consisted of individuals diagnosed with peri-implant health, peri-implant mucositis, or peri-implantitis, classified according to clinical and radiographic findings. All participants provided informed consent before sample collection.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
HIF-1α, GPX-4, and MDA Levels in Peri-Implant Crevicular Fluid | Cross-sectional measurement at a single time point
  Measurement of hypoxia-inducible factor-1 alpha (HIF-1α), glutathione peroxidase-4 (GPX-4), and malondialdehyde (MDA) levels in peri-implant crevicular fluid using enzyme-linked immunosorbent assay (ELISA) to assess their association with peri-implant health, mucositis, and peri-implantitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Faculty of Dentistry, Department of Periodontology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding individual participant data (IPD) sharing has not yet been finalized. Factors such as data privacy regulations, institutional policies, and publication plans will be considered before determining whether and to what extent the collected IPD will be shared.

REFERENCES:
- [Result] Gao X, Hu W, Qian D, Bai X, He H, Li L, Sun S. The Mechanisms of Ferroptosis Under Hypoxia. Cell Mol Neurobiol. 2023 Oct;43(7):3329-3341. doi: 10.1007/s10571-023-01388-8. Epub 2023 Jul 17. PMID 37458878
- [Result] Hsieh CH, Lin YJ, Chen WL, Huang YC, Chang CW, Cheng FC, Liu RS, Shyu WC. HIF-1alpha triggers long-lasting glutamate excitotoxicity via system xc- in cerebral ischaemia-reperfusion. J Pathol. 2017 Feb;241(3):337-349. doi: 10.1002/path.4838. Epub 2016 Dec 29. PMID 27801527
- [Result] Fan Y, Ma L, Fang X, Du S, Mauck J, Loor JJ, Sun X, Jia H, Xu C, Xu Q. Role of hypoxia-inducible-factor-1alpha (HIF-1alpha) in ferroptosis of adipose tissue during ketosis. J Dairy Sci. 2024 Dec;107(12):10611-10627. doi: 10.3168/jds.2024-24822. Epub 2024 Jul 26. PMID 39067746
- [Result] Afacan B, Ozturk VO, Pasali C, Bozkurt E, Kose T, Emingil G. Gingival crevicular fluid and salivary HIF-1alpha, VEGF, and TNF-alpha levels in periodontal health and disease. J Periodontol. 2019 Jul;90(7):788-797. doi: 10.1002/JPER.18-0412. Epub 2018 Dec 11. PMID 30536725
- [Result] Xing L, Dong W, Chen Y, Dai W, Xiao X, Liu Z, Zhang X, Bai D, Xu H. Fibroblast ferroptosis is involved in periodontitis-induced tissue damage and bone loss. Int Immunopharmacol. 2023 Jan;114:109607. doi: 10.1016/j.intimp.2022.109607. Epub 2022 Dec 22. PMID 36700777
- [Result] Qiao S, Li B, Cai Q, Li Z, Yin Z, He J, Li Y, Meng W. Involvement of ferroptosis in Porphyromonas gingivalis lipopolysaccharide-stimulated periodontitis in vitro and in vivo. Oral Dis. 2023 Nov;29(8):3571-3582. doi: 10.1111/odi.14292. Epub 2022 Jul 12. PMID 35765229